CLINICAL TRIAL: NCT01595867
Title: A Randomized, Double-Blind, Placebo-Controlled, 3 Way Crossover Study Evaluating The Relative Abuse Potential Of Crushed Embeda Compared To Morphine Sulfate Controlled Release Tablets (Crushed) And Placebo In Non-Dependent, Recreational Opioid Users Following Intranasal Administration
Brief Title: Abuse Potential Assessment of Intranasally Administered EMBEDA Compared To Morphine Sulfate Controlled Release And Placebo
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: ALO-01-10-4004; B4541005
Record Dates: First submitted 2012-05-08; First posted 2012-05-10 (Estimated); Last update posted 2012-06-08 (Estimated); Status verified 2012-06

CONDITIONS: Narcotic Abuse; Opioid-related Disorders; Analgesia; Chronic Pain
Keywords: abuse liability; abuse potential; morphine; intranasal administration; snorting; opioid abuse; pharmacodynamic; recreational drug use
MeSH Terms: conditions — Narcotic-Related Disorders; Opioid-Related Disorders; Agnosia; Chronic Pain; Recreational Drug Use | interventions — Naltrexone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treatment A (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- Treatment B (Experimental): EMBEDA 30 mg crushed
  Interventions: Drug: EMBEDA - morphine sulfate/ naltrexone hydrochloride
- Treatment C (Active Comparator): Morphine Sulfate Controlled Release 30 mg crushed
  Interventions: Drug: morphine sulfate CR crushed.

INTERVENTIONS:
Drug: Placebo — Lactose (100 mg) placebo tablets crushed; single dose
  Arms: Treatment A
Drug: EMBEDA - morphine sulfate/ naltrexone hydrochloride — EMBEDA (morphine sulfate/naltrexone hydrochloride) 30 mg/ 1.2 mg extended release; capsule contents crushed; single dose
  Arms: Treatment B
Drug: morphine sulfate CR crushed. — Morphine sulfate controlled release 30 mg tablet crushed
  Arms: Treatment C

SUMMARY:
This was a single-dose, randomized, double-blind, placebo-controlled, 3 way crossover study designed to evaluate the relative abuse potential of crushed EMBEDA® compared to morphine sulfate CR tablets and placebo in healthy male and female, non-dependent, recreational opioid users. An appropriate dose of morphine sulfate CR (i.e., 30 mg, 60 or 90 mg) was to be selected during Part A of the study (Dose Selection Phase). Each subject participated in the study for up to (approximately) 16 weeks and was confined in the clinic for a total of up to 12 nights.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subjects 18 to 55 years of age, inclusive.
* Subject is a recreational opioid user who is NOT dependent on opioids based on Diagnostic and Statistical Manual of Mental Disorders-Fourth Edition-Text Revision (DSM-IV-TR) criteria and the Naloxone Challenge. A recreational opioid user is defined as use of opioids for non-therapeutic purposes (i.e., for psychoactive effects) on at least 10 occasions within the last year and at least once in the 12 weeks before the Screening Visit (Visit 1).
* Subjects must have experience with intranasal drug administration, defined as intranasal use on at least 3 occasions within the last year prior to the Screening Visit.

Exclusion Criteria:

* Diagnosis of substance and/or alcohol dependence (excluding caffeine and nicotine), as assessed by the Investigator using the DSM IV-TR criteria.
* Has participated in, is currently participating in, or is seeking treatment for substance- and or alcohol-related disorders (excluding nicotine and caffeine).
* Has any condition in which an opioid is contraindicated; e.g., significant respiratory depression, acute or severe bronchial asthma or hypercarbia, or is suspected of having paralytic ileus.
* Allergy or history of hypersensitivity to morphine sulfate, other opioids, naltrexone hydrochloride, naloxone, and/or lactose.
* History or current clinically significant neurological, cardiovascular, renal, hepatic, endocrine, gastrointestinal, hematologic, or metabolic disease as evaluated by the Investigator.
* History or current pulmonary disease including asthma, chronic obstructive pulmonary disease, exercise-induced asthma, bronchitis, and obstructive sleep apnea.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2010-08; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Drug Liking Visual Analog Scale maximum peak effect (Emax) | 0.5, 1, 1.5, 2, 3, 4, 6, 8,12, and 24 hours post-dose
Drug Liking Visual Analog Scale Area under the effect curve to 2 hours (AUE0-2h) | 0.5, 1, 1.5, 2, 3, 4, 6, 8,12, and 24 hours post-dose
High Visual Analog Scale maximum peak effect (Emax) | pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8,12, and 24 hours post-dose
High Visual Analog Scale Area under the effect curve to 2 hours (AUE0-2h) | pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8,12, and 24 hours post-dose

SECONDARY OUTCOMES:
Drug Liking Visual Analog Scale Area under the effect curve to 1 hour (AUE0-1h) | 0.5, 1, 1.5, 2, 3, 4, 6, 8,12, and 24 hours post-dose
Drug Liking Visual Analog Scale Area under the effect curve to 4 hours (AUE0-4h) | 0.5, 1, 1.5, 2, 3, 4, 6, 8,12, and 24 hours post-dose
Drug Liking Visual Analog Scale Area under the effect curve to 8 hours (AUE0-8h) | 0.5, 1, 1.5, 2, 3, 4, 6, 8,12, and 24 hours post-dose
Drug Liking Visual Analog Scale Area under the effect curve to 12 hours (AUE0-12h) | 0.5, 1, 1.5, 2, 3, 4, 6, 8,12, and 24 hours post-dose
Drug Liking Visual Analog Scale Area under the effect curve to 24 hours (AUE0-24h) | 0.5, 1, 1.5, 2, 3, 4, 6, 8,12, and 24 hours post-dose
Drug Liking Visual Analog Scale Area time to maximum effect (TEmax) | 0.5, 1, 1.5, 2, 3, 4, 6, 8,12, and 24 hours post-dose
High VVisual Analog Scale Area under the effect curve to 1 hour (AUE0-1h) | pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8,12, and 24 hours post-dose
High Visual Analog Scale Area under the effect curve to 4 hours (AUE0-4h) | pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8,12, and 24 hours post-dose
High Visual Analog Scale Area under the effect curve to 8 hours (AUE0-8h) | pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8,12, and 24 hours post-dose
High Visual Analog Scale Area under the effect curve to 12 hours (AUE0-12h) | pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8,12, and 24 hours post-dose
High Visual Analog Scale Area under the effect curve to 24 hours (AUE0-24h) | pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8,12, and 24 hours post-dose
High Visual Analog Scale Area time to maximum effect (TEmax) | pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8,12, and 24 hours post-dose
Any Drug Effects Visual Analog Scale maximum peak effect (Emax) | 0.5, 1, 1.5, 2, 3, 4, 6, 8,12, and 24 hours post-dose
Any Drug Effects Visual Analog Scale Area under the effect curve to 2 hours (AUE0-2h) | 0.5, 1, 1.5, 2, 3, 4, 6, 8,12, and 24 hours post-dose
Any Drug Effects Visual Analog Scale Area under the effect curve to 1 hour (AUE0-1h) | 0.5, 1, 1.5, 2, 3, 4, 6, 8,12, and 24 hours post-dose
Any Drug Effects Visual Analog Scale Area under the effect curve to 4 hours (AUE0-4h) | 0.5, 1, 1.5, 2, 3, 4, 6, 8,12, and 24 hours post-dose
Any Drug Effects Visual Analog Scale Area under the effect curve to 8 hours (AUE0-8h) | 0.5, 1, 1.5, 2, 3, 4, 6, 8,12, and 24 hours post-dose
Any Drug Effects Visual Analog Scale Area under the effect curve to 12 hours (AUE0-12h) | 0.5, 1, 1.5, 2, 3, 4, 6, 8,12, and 24 hours post-dose
Any Drug Effects Visual Analog Scale Area under the effect curve to 24 hours (AUE0-24h) | 0.5, 1, 1.5, 2, 3, 4, 6, 8,12, and 24 hours post-dose
Any Drug Effects Visual Analog Scale Area time to maximum effect (TEmax) | 0.5, 1, 1.5, 2, 3, 4, 6, 8,12, and 24 hours post-dose
Good Drug Effects Visual Analog Scale maximum peak effect (Emax) | 0.5, 1, 1.5, 2, 3, 4, 6, 8,12, and 24 hours post-dose
Good Drug Effects Visual Analog Scale Area under the effect curve to 1 hour (AUE0-1h) | 0.5, 1, 1.5, 2, 3, 4, 6, 8,12, and 24 hours post-dose
Good Drug Effects Visual Analog Scale Area under the effect curve to 2 hours (AUE0-2h) | 0.5, 1, 1.5, 2, 3, 4, 6, 8,12, and 24 hours post-dose
Good Drug Effects Visual Analog Scale Area under the effect curve to 4 hours (AUE0-4h) | 0.5, 1, 1.5, 2, 3, 4, 6, 8,12, and 24 hours post-dose
Good Drug Effects Visual Analog Scale Area under the effect curve to 8 hours (AUE0-8h) | 0.5, 1, 1.5, 2, 3, 4, 6, 8,12, and 24 hours post-dose
Good Drug Effects Visual Analog Scale Area under the effect curve to 12 hours (AUE0-12h) | 0.5, 1, 1.5, 2, 3, 4, 6, 8,12, and 24 hours post-dose
Good Drug Effects Visual Analog Scale Area under the effect curve to 24 hours (AUE0-24h) | 0.5, 1, 1.5, 2, 3, 4, 6, 8,12, and 24 hours post-dose
Good Drug Effects Visual Analog Scale Area time to maximum effect (TEmax) | 0.5, 1, 1.5, 2, 3, 4, 6, 8,12, and 24 hours post-dose
Bad Drug Effects Visual Analog Scale maximum peak effect (Emax) | 0.5, 1, 1.5, 2, 3, 4, 6, 8,12, and 24 hours post-dose
Bad Drug Effects Visual Analog Scale Area under the effect curve to 1 hour (AUE0-1h) | 0.5, 1, 1.5, 2, 3, 4, 6, 8,12, and 24 hours post-dose
Bad Drug Effects Visual Analog Scale Area under the effect curve to 2 hours (AUE0-2h) | 0.5, 1, 1.5, 2, 3, 4, 6, 8,12, and 24 hours post-dose
Bad Drug Effects Visual Analog Scale Area under the effect curve to 4 hours (AUE0-4h) | 0.5, 1, 1.5, 2, 3, 4, 6, 8,12, and 24 hours post-dose
Bad Drug Effects Visual Analog Scale Area under the effect curve to 8 hours (AUE0-8h) | 0.5, 1, 1.5, 2, 3, 4, 6, 8,12, and 24 hours post-dose
Bad Drug Effects Visual Analog Scale Area under the effect curve to 12 hours (AUE0-12h) | 0.5, 1, 1.5, 2, 3, 4, 6, 8,12, and 24 hours post-dose
Bad Drug Effects Visual Analog Scale Area under the effect curve to 24 hours (AUE0-24h) | 0.5, 1, 1.5, 2, 3, 4, 6, 8,12, and 24 hours post-dose
Bad Drug Effects Visual Analog Scale Area time to maximum effect (TEmax) | 0.5, 1, 1.5, 2, 3, 4, 6, 8,12, and 24 hours post-dose
Feel Sick Visual Analog Scale maximum peak effect (Emax) | pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8,12, and 24 hours post-dose
Feel Sick Visual Analog Scale Area under the effect curve to 1 hour (AUE0-1h) | pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8,12, and 24 hours post-dose
Feel Sick Visual Analog Scale Area under the effect curve to 2 hours (AUE0-2h) | pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8,12, and 24 hours post-dose
Feel Sick Visual Analog Scale Area under the effect curve to 4 hours (AUE0-4h) | pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8,12, and 24 hours post-dose
Feel Sick Visual Analog Scale Area under the effect curve to 8 hours (AUE0-8h) | pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8,12, and 24 hours post-dose
Feel Sick Visual Analog Scale Area under the effect curve to 12 hours (AUE0-12h) | pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8,12, and 24 hours post-dose
Feel Sick Visual Analog Scale Area under the effect curve to 24 hours (AUE0-24h) | pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8,12, and 24 hours post-dose
Feel Sick Visual Analog Scale Area time to maximum effect (TEmax) | pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8,12, and 24 hours post-dose
Nausea Visual Analog Scale maximum peak effect (Emax) | pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8,12, and 24 hours post-dose
Nausea Visual Analog Scale Area under the effect curve to 1 hour (AUE0-1h) | pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8,12, and 24 hours post-dose
Nausea Visual Analog Scale Area under the effect curve to 2 hours (AUE0-2h) | pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8,12, and 24 hours post-dose
Nausea Visual Analog Scale Area under the effect curve to 4 hours (AUE0-4h) | pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8,12, and 24 hours post-dose
Nausea Visual Analog Scale Area under the effect curve to 8 hours (AUE0-8h) | pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8,12, and 24 hours post-dose
Nausea Visual Analog Scale Area under the effect curve to 12 hours (AUE0-12h) | pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8,12, and 24 hours post-dose
Nausea Visual Analog Scale Area under the effect curve to 24 hours (AUE0-24h) | pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8,12, and 24 hours post-dose
Nausea Visual Analog Scale Area time to maximum effect (TEmax) | pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8,12, and 24 hours post-dose
Sleepy Visual Analog Scale maximum peak effect (Emax) | pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8,12, and 24 hours post-dose
Sleepy Visual Analog Scale Area under the effect curve to 1 hour (AUE0-1h) | pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8,12, and 24 hours post-dose
Sleepy Visual Analog Scale Area under the effect curve to 2 hours (AUE0-2h) | pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8,12, and 24 hours post-dose
Sleepy Visual Analog Scale Area under the effect curve to 4 hours (AUE0-4h) | pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8,12, and 24 hours post-dose
Sleepy Visual Analog Scale Area under the effect curve to 8 hours (AUE0-8h) | pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8,12, and 24 hours post-dose
Sleepy Visual Analog Scale Area under the effect curve to 12 hours (AUE0-12h) | pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8,12, and 24 hours post-dose
Sleepy Visual Analog Scale Area under the effect curve to 24 hours (AUE0-24h) | pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8,12, and 24 hours post-dose
Sleepy Visual Analog Scale Area time to maximum effect (TEmax) | pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8,12, and 24 hours post-dose
Dizzy Visual Analog Scale maximum peak effect (Emax) | pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8,12, and 24 hours post-dose
Dizzy Visual Analog Scale Area under the effect curve to 1 hour (AUE0-1h) | pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8,12, and 24 hours post-dose
Dizzy Visual Analog Scale Area under the effect curve to 2 hours (AUE0-2h) | pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8,12, and 24 hours post-dose
Dizzy Visual Analog Scale Area under the effect curve to 4 hours (AUE0-4h) | pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8,12, and 24 hours post-dose
Dizzy Visual Analog Scale Area under the effect curve to 8 hours (AUE0-8h) | pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8,12, and 24 hours post-dose
Dizzy Visual Analog Scale Area under the effect curve to 12 hours (AUE0-12h) | pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8,12, and 24 hours post-dose
Dizzy Visual Analog Scale Area under the effect curve to 24 hours (AUE0-24h) | pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8,12, and 24 hours post-dose
Dizzy Visual Analog Scale Area time to maximum effect (TEmax) | pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8,12, and 24 hours post-dose
Pupil Diameter minimum peak effect (Emin) | pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8,12, and 24 hours post-dose
Pupil Diameter time to minimum peak effect (TEmin) | pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8,12, and 24 hours post-dose
Pupil Diameter Area under the effect curve to 1 hour (AUE0-1h) | pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8,12, and 24 hours post-dose
Pupil Diameter Area under the effect curve to 2 hours (AUE0-2h) | pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8,12, and 24 hours post-dose
Pupil Diameter Area under the effect curve to 4 hours (AUE0-4h) | pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8,12, and 24 hours post-dose
Pupil Diameter Area under the effect curve to 8 hours (AUE0-8h) | pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8,12, and 24 hours post-dose
Pupil Diameter Area under the effect curve to 12 hours (AUE0-12h) | pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8,12, and 24 hours post-dose
Pupil Diameter Area under the effect curve to 24 hours (AUE0-24h) | pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8,12, and 24 hours post-dose
Take Drug Again Visual Analog Scale maximum peak effect (Emax) | 12 and 24 hours post dose
Take Drug Again Visual Analog Scale mean (Emean) | 12 and 24 hours post dose
Overall Drug Liking Visual Analog Scale maximum peak effect (Emax) | 12 and 24 hours post dose
Overall Drug Liking Visual Analog Scale mean (Emean) | 12 and 24 hours post dose
Subject Rating Scale - Need to Blow Nose maximum peak effect (Emax) | pre dose and 0.5, 1, 1.5, and 2 hours post dose
Subject Rating Scale - Need to Blow Nose Area under the effect curve to 1 hour (AUE0-1h) | pre dose and 0.5, 1, 1.5, and 2 hours post dose
Subject Rating Scale - Need to Blow Nose Area under the effect curve to 2 hours (AUE0-2h) | pre dose and 0.5, 1, 1.5, and 2 hours post dose
Subject Rating Scale - Runny Nose/Nasal Discharge maximum peak effect (Emax) | pre dose and 0.5, 1, 1.5, and 2 hours post dose
Subject Rating Scale - Runny Nose/Nasal Discharge Area under the effect curve to 1 hour (AUE0-1h) | pre dose and 0.5, 1, 1.5, and 2 hours post dose
Subject Rating Scale - Runny Nose/Nasal Discharge Area under the effect curve to 2 hours (AUE0-2h) | pre dose and 0.5, 1, 1.5, and 2 hours post dose
Subject Rating Scale - Burning maximum peak effect (Emax) | pre dose and 0.5, 1, 1.5, and 2 hours post dose
Subject Rating Scale - Burning Area under the effect curve to 1 hour (AUE0-1h) | pre dose and 0.5, 1, 1.5, and 2 hours post dose
Subject Rating Scale - Burning Area under the effect curve to 2 hours (AUE0-2h) | pre dose and 0.5, 1, 1.5, and 2 hours post dose
Subject Rating Scale - Facial Pain/Pressure maximum peak effect (Emax) | pre dose and 0.5, 1, 1.5, and 2 hours post dose
Subject Rating Scale - Facial Pain/Pressure Area under the effect curve to 1 hour (AUE0-1h) | pre dose and 0.5, 1, 1.5, and 2 hours post dose
Subject Rating Scale - Facial Pain/Pressure Area under the effect curve to 2 hours (AUE0-2h) | pre dose and 0.5, 1, 1.5, and 2 hours post dose
Subject Rating Scale - Nasal Congestion maximum peak effect (Emax) | pre dose and 0.5, 1, 1.5, and 2 hours post dose
Subject Rating Scale - Nasal Congestion Area under the effect curve to 1 hour (AUE0-1h) | pre dose and 0.5, 1, 1.5, and 2 hours post dose
Subject Rating Scale - Nasal Congestion Area under the effect curve to 2 hours (AUE0-2h) | pre dose and 0.5, 1, 1.5, and 2 hours post dose
Plasma morphine - Maximum observed plasma concentration (Cmax) | pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours post-dose
Plasma morphine - Time to maximum observed plasma concentration (Tmax) | pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours post-dose
Plasma morphine - Area under the plasma concentration time curve from time zero to 1 hour (AUC0-1h) | pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours post-dose
Plasma morphine - Area under the plasma concentration time curve from time zero to 2 hours (AUC0-2h) | pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours post-dose
Plasma morphine - Area under the plasma concentration time curve from time zero to 4 hours (AUC0-4h) | pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours post-dose
Plasma 6-ß-naltrexol - Maximum observed plasma concentration (Cmax) | pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours post-dose
Plasma 6-ß-naltrexol - Area under the plasma concentration time curve from time zero to 1 hour (AUC0-1h) | pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours post-dose
Plasma 6-ß-naltrexol - Area under the plasma concentration time curve from time zero to 12 hours (AUC0-12h) | pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours post-dose
Plasma 6-ß-naltrexol - Area under the plasma concentration time curve from time zero to 24 hours (AUC0-24h) | pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours post-dose
Plasma 6-ß-naltrexol - Area under the plasma concentration time curve from time zero to 4 hours (AUC0-4h) | pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours post-dose
Plasma 6-ß-naltrexol - Area under the plasma concentration time curve from time zero to 8 hours (AUC0-8h) | pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours post-dose
Plasma 6-ß-naltrexol - Time to maximum observed plasma concentration (Tmax | pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours post-dose
Plasma 6-ß-naltrexol- Area under the plasma concentration time curve from time zero to 2 hours (AUC0-2h) | pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours post-dose
Plasma 6-ß-naltrexol- Area under the plasma concentration time curve from time zero to infinity (AUC0-8), as applicable | pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours post-dose
Plasma morphine - Area under the plasma concentration time curve from time zero to 12 hours (AUC0-12h) | pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours post-dose
Plasma morphine - Area under the plasma concentration time curve from time zero to 24 hours (AUC0-24h) | pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours post-dose
Plasma morphine - Area under the plasma concentration time curve from time zero to 8 hours (AUC0-8h) | pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours post-dose
Plasma morphine - Area under the plasma concentration time curve from time zero to infinity (AUC0-8), as applicable | pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours post-dose
Plasma naltrexone - Area under the plasma concentration time curve from time zero to 1 hour (AUC0-1h) | pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours post-dose
Plasma naltrexone - Area under the plasma concentration time curve from time zero to 12 hours (AUC0-12h) | pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours post-dose
Plasma naltrexone - Area under the plasma concentration time curve from time zero to 24 hours (AUC0-24h) | pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours post-dose
Plasma naltrexone - Area under the plasma concentration time curve from time zero to 4 hours (AUC0-4h) | pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours post-dose
Plasma naltrexone - Area under the plasma concentration time curve from time zero to 8 hours (AUC0-8h) | pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours post-dose
Plasma naltrexone - Area under the plasma concentration time curve from time zero to infinity (AUC0-8), as applicable | pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours post-dose
Plasma naltrexone - Maximum observed plasma concentration (Cmax) | pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours post-dose
Plasma naltrexone - Time to maximum observed plasma concentration (Tmax) | pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours post-dose
Plasma naltrexone- Area under the plasma concentration time curve from time zero to 2 hours (AUC0-2h) | pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- [Derived] Setnik B, Goli V, Levy-Cooperman N, Mills C, Shram M, Smith I. Assessing the subjective and physiological effects of intranasally administered crushed extended-release morphine formulations with and without a sequestered naltrexone core in recreational opioid users. Pain Res Manag. 2013 Jul-Aug;18(4):e55-62. doi: 10.1155/2013/952082. PMID 23936895
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=ALO-01-10-4004&StudyName=Abuse%20Potential%20Assessment%20of%20Intranasally%20Administered%20EMBEDA%20Compared%20To%20Morphine%20Sulfate%20Controlled%20Release%20And%20Placebo%20